CLINICAL TRIAL: NCT01789606
Title: Ibuprofen 600 Mg Immediate Release/Extended Release (IR/ER) Caplet Self-selection, Safety And Compliance Study
Brief Title: Self-Selection and Actual Use Trial of Ibuprofen 600 mg Immediate Release/Extended Caplet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4371008; AK-10-11 (Other: Alias Study Number)
Record Dates: First submitted 2012-09-19; First posted 2013-02-12 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Analgesia
Keywords: Self-selection and actual use/compliance trial.
MeSH Terms: conditions — Agnosia | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibuprofen 600 mg Immediate Release/Extended Release Caplet (Experimental)
  Interventions: Drug: Ibuprofen 600 mg Immediate Release/Extended Release Caplet

INTERVENTIONS:
Drug: Ibuprofen 600 mg Immediate Release/Extended Release Caplet — Ibuprofen 600 mg Immediate Release/Extended Release Caplet to be adminstered orally (i.e., one caplet every 12 hours, not to exceed 2 caplets per day) for pain.

SUMMARY:
A self-selection and actual use trial to evaluate the extent to which consumers will appropriately select and use the 600 mg immediate release/extended release caplets and comply with dosing instructions.

ELIGIBILITY:
Inclusion Criteria:

* at least 12 years of age
* use of at least 5 doses per month of over-the-counter pain relievers over the past 3 months
* provide written informed consent (subjects 12-<18 years of age provide a written assent and parent/guardian will provide written informed consent)
* capable of and willing to swallow the study medication

Exclusion Criteria:

* participated in other research studies in the last 6 months
* they or someone else in their household work for a pharmaceutical company, is a relative of study site personnel involved with the study, or an immediate family member is already enrolled in the study
* have a history of known allergies to ibuprofen, aspirin, or other NSAIDs
* have a history of heart surgery in the last 60 days or planned heart surgery in the next 60 days
* female subjects are pregnant or breast feeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1083 (Actual)
Dates: Start 2012-09-24 (Actual); Primary Completion 2013-06-03 (Actual); Study Completion 2013-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Medical Arts Rexall Pharmacy, Anaheim, California
  - B and B Pharmacy, Yorba Linda, California
  - Wynn's Pharmacy Inc., Griffin, Georgia
  - Stark Pharmacy, Overland Park, Kansas
  - Catonsville Pharmacy, Baltimore, Maryland
  - Goodrich Pharmacy, Blaine, Minnesota
  - Kemper Drug, Elk River, Minnesota
  - Cub Pharmacy Number 1924, Saint Louis Park, Minnesota
  - Albers' Medical Pharmacy, Kansas City, Missouri
  - Countryside Pharmacy, Savannah, Missouri
  - Duran Central Pharmacy, Albuquerque, New Mexico
  - Total Health and Wellness Center of Taos, Taos, New Mexico
  - The Medicine Shoppe, Ogden, Utah
  - The Medicine Shoppe, Salt Lake City, Utah
  - Family Plaza Pharmacy, West Jordan, Utah
  - Montpelier Pharmacy, Inc., Montpelier, Virginia
  - Ostrom Drugs, Kenmore, Washington
  - Kusler's Pharmacy, Snohomish, Washington

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Paluch E, Jayawardena S, Wilson B, Farnsworth S. Consumer self-selection, safety, and compliance with a novel over-the-counter ibuprofen 600-mg immediate-release and extended-release tablet. J Am Pharm Assoc (2003). 2016 Jul-Aug;56(4):397-404. doi: 10.1016/j.japh.2016.03.003. Epub 2016 May 13. PMID 27184785
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4371008&StudyName=Self-Selection%20and%20Actual%20Use%20Trial%20of%20Ibuprofen%20600%20mg%20Immediate%20Release/Extended%20Caplet

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-Selection Arm: Participants who were enrolled in the self-selection arm and completed the self-selection questionnaire were made to either select or deselect Ibuprofen 200 milligram (mg) immediate release (IR) or 600 mg IR or extended release (ER) tablets, or to deselect both the products based on their current painful condition. Participants enrolled in this arm did not receive any study medication.
- Compliance Arm: Participants enrolled in compliance arm, received at least one dose of 600 mg IR or ER tablet of Ibuprofen over a period of 30 days and returned the diary cards, or if any information on dosing was available.
Period: Overall Study
Arm/Group | Self-Selection Arm | Compliance Arm
Started | 251 | 832
Completed | 228 | 382
Not Completed | 23 | 450
Not completed — Participant not Purchased the Product | 0 | 20
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Ineligible | 6 | 2
Not completed — Administrative Reasons | 17 | 6
Not completed — No Study Medication Taken | 0 | 1
Not completed — Protocol Violation | 0 | 55
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 0 | 14
Not completed — Ineligible or not Willing to Continue | 0 | 348

BASELINE CHARACTERISTICS:
Population: Analysis population included all the participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Selection Arm | Compliance Arm | Total
Number analyzed (Participants) | 251 | 832 | 1083
Age, Customized [Number; unit: participants]
  Less Than (<)18 years | 2 | 5 | 7
  Greater Than or Equal to (>=) 18 years | 247 | 827 | 1074
  Unknown | 2 | 0 | 2
Sex/Gender, Customized [Number; unit: participants]
  Female | 114 | 408 | 522
  Male | 114 | 403 | 517
  Unknown | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Correctly Select to Use or Correctly De-select Not to Use Ibuprofen 600 Milligram (mg) Immediate Release (IR) or Extended Release (ER) Study Medication
Description: Participants as correct selectors included all participants who selected Ibuprofen 600 mg IR/ER medication with the last episode of pain of >=6 hours, if left untreated. Participants as correct de-selectors included all participants who either selected Ibuprofen 200 mg or selected 'neither' with a typical pain duration of less than (<) 6 hours, if left untreated.
Time Frame: Day 1
Population: This outcome measure was not planned to be analysed in compliance arm. Analysis population included all participants enrolled in the self-selection arm of the study and completed the self-selection questionnaire.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Self-Selection Arm
Number analyzed (Participants) | 249
percentage of participants | 69.1 [63.3 to 74.8]

2. Primary Outcome: Percentage of Participants Who Correctly Select to Use or Correctly De-select Not to Use Ibuprofen 600 mg IR/ER Study Medication Excluding Those Classified as Missed Opportunity
Description: Participants as correct selectors included all participants who selected Ibuprofen 600 mg IR/ER medication with the last episode of pain of >=6 hours, if left untreated. Participants as correct de-selectors included all participants who either selected Ibuprofen 200 mg or selected 'neither' with a typical pain duration of <6 hours, if left untreated. Participants were classified as "missed opportunity" cases when they selected the Ibuprofen 200 mg IR medication with their typical duration of pain >=6 hours.
Time Frame: Day 1
Population: This outcome measure was not planned to be analysed in compliance arm. Analysis population included all participants enrolled in the self-selection arm of the study and completed the self-selection questionnaire. Here, 'Number of Participants Analyzed (N)' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Self-Selection Arm
Number analyzed (Participants) | 208
percentage of participants | 82.7 [77.6 to 87.8]

3. Primary Outcome: Percentage of Participants Who Select to Use Ibuprofen 600 mg IR/ER Medication With a Typical Pain Duration of Less Than (<) 6 Hours
Description: Percentage of participants with correct selection of Ibuprofen 600 mg IR/ER medication with a typical duration of pain <6 hours were reported in this outcome measure.
Time Frame: Day 1
Population: This outcome measure was not planned to be analysed in compliance arm. Analysis population included all participants enrolled in the self-selection arm of the study and completed the self-selection questionnaire. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Self-Selection Arm
Number analyzed (Participants) | 38
percentage of participants | 63.2 [47.8 to 78.5]

4. Primary Outcome: Percentage of Participants Who Select to Use Ibuprofen 200 mg IR Medication With a Typical Pain Duration of Greater Than or Equal to (>=) 6 Hours
Description: Percentage of participants with selection of Ibuprofen 200 mg IR medication with a typical duration of pain >=6 hours were reported in this outcome measure. These participants were classified as ''missed opportunity'' cases.
Time Frame: Day 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Self-Selection Arm
Number analyzed (Participants) | 211
percentage of participants | 20.9 [15.4 to 26.3]

5. Primary Outcome: Percentage of Participants With the Use of Study Medication For Greater Than (>) 10 Days With an Average Daily Dose of Greater Than (>) 1600 mg
Description: Percentage of participants with the use of study medication for >10 days with an average daily dose of >1600 mg were reported in this outcome measure.
Time Frame: Day 1 up to Day 30
Population: This outcome measure was not planned to be analysed in self-selection arm. Analysis population included all participants of compliance arm who received at least 1 dose of the study drug during the 30 days and returned the completed study diary, or any information on dosing which was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Compliance Arm
Number analyzed (Participants) | 403
percentage of participants | 1.2 [0.2 to 2.3]

6. Primary Outcome: Percentage of Participants With the Use of Study Medication For Less Than or Equal to (<=) 10 Days and Use More Than 20 Tablets With an Average Daily Dose of Greater Than (>) 1600 mg
Description: Percentage of participants who used the study medication for <=10 days and used more than 20 tablets with an average daily dose of >1600 mg were reported in this outcome measure.
Time Frame: Day 1 up to Day 30
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Compliance Arm
Number analyzed (Participants) | 403
percentage of participants | 0 [0 to 0]

7. Secondary Outcome: Average Daily Dose Among Excessive Users
Description: Excessive users included all participants who used the study medication for more than 10 days (not necessarily consecutive) during study period with an average daily dose of >1600 mg or all participants who used the study medication for <=10 days during study period, used more than 20 tablets and had an average daily dose of >1600 mg.
Time Frame: Day 1 up to Day 30
Population: This outcome measure was not planned to be analysed in self-selection arm. Analysis population included all participants of compliance arm who received at least 1 dose of the study drug during the 30 days and returned the completed study diary, or any information on dosing which was available. 'N' is participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Compliance Arm
Number analyzed (Participants) | 5
milligram | 1821.1 (157.4)

8. Secondary Outcome: Number of Dosing Days Among Inappropriate Users
Description: Participants were considered as inappropriate users if they improperly used the study medication in their last pain episode duration of <6 hours, if left untreated, based on the information provided at the follow up interview.
Time Frame: Day 1 up to Day 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Compliance Arm
Number analyzed (Participants) | 45
days | 14.8 (8.1)

9. Secondary Outcome: Number of Pain Episodes Treated With Single Dose or Multiple Dose Among Inappropriate Users
Description: In this outcome measure, number of pain episodes treated with single dose or multiple dose per day among inappropriate users were reported. Participants were considered as inappropriate users if they improperly used the study medication in their last pain episode duration of <6 hours, based on the information provided at the follow up interview.
Time Frame: Day 1 up to Day 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pain episodes
Arm/Group | Compliance Arm
Number analyzed (Participants) | 45
pain episodes
  Single dose | 13.1 (7.4)
  Multiple dose | 1.8 (2.6)

10. Secondary Outcome: Number of Treatment Days Exceeding the Daily Dose of 1200 Milligram
Description: Number of treatment days when participants exceeded the daily dose of 1200 milligram were reported in this outcome measure.
Time Frame: Day 1 up to Day 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Compliance Arm
Number analyzed (Participants) | 403
days | 0.31 (1.188)

11. Secondary Outcome: Number of Treatment Days Exceeding the Daily Dose of 1200 Milligram Excluding Treatment of Severe Symptoms
Description: In this outcome measure, number of treatment days exceeding the daily dose of 1200 mg, excluding the days when severe symptoms were treated, were reported.
Time Frame: Day 1 up to Day 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Compliance Arm
Number analyzed (Participants) | 403
days | 0.12 (0.637)

12. Secondary Outcome: Number of Dosing Occasions Exceeding the Single Dose of 600 Milligram
Description: In this outcome measure, number of dosing occasions exceeding the single dose of 600 mg were reported.
Time Frame: Day 1 up to Day 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: dosing occasions
Arm/Group | Compliance Arm
Number analyzed (Participants) | 403
dosing occasions | 1.48 (4.185)

13. Secondary Outcome: Number of Dosing Occasions Exceeding the Single Dose of 600 Milligram Excluding Treatment of Severe Symptoms
Description: In this outcome measure, number of dosing occasions exceeding the single dose of 600 mg, excluding the events when severe symptoms were treated, were reported.
Time Frame: Day 1 up to Day 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: dosing occasions
Arm/Group | Compliance Arm
Number analyzed (Participants) | 403
dosing occasions | 0.83 (3.020)

14. Secondary Outcome: Average Daily Dose of Study Medication
Time Frame: Day 1 up to Day 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Compliance Arm
Number analyzed (Participants) | 403
milligram | 781.0 (229.3)

15. Secondary Outcome: Maximum Daily Dose of Study Medication
Time Frame: Day 1 up to Day 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Compliance Arm
Number analyzed (Participants) | 403
milligram | 1147.9 (604.43)

ADVERSE EVENTS:
Description: Safety data collected for all participants who received at least 1 dose of study drug(safety population).Same event may appear as AE and SAE.However,distinct events are presented.An event may categorized as serious in 1 participant and as nonserious in other participant,or 1 participant may experience both serious and nonserious event during study.
Arm/Group | Compliance Arm
Serious Adverse Events (participants affected / at risk) | 1/405
Other Adverse Events (participants affected / at risk) | 163/405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Compliance Arm (N=405)
Pleural infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Compliance Arm (N=405)
Ear pain (Ear and labyrinth disorders) | 2
Vision blurred (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 26
Chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 3
Diverticulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 59
Pharyngitis streptococcal (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 6
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Animal bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 6
Limb injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 15
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Hypoaesthesia (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 2
Tension headache (Nervous system disorders) | 6
Renal pain (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1/223 — This is gender specific event. The number of participants evaluable for this event are 223.
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Rosacea (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.